CLINICAL TRIAL: NCT06752122
Title: Safety, Tolerability and Pharmacokinetics of Single-ascending Doses of RCS-21 in Healthy Volunteers. A Double Blind, Randomized, Placebo Controlled Phase I Study.
Brief Title: Safety, Tolerability, and Pharmacokinetics of RCS-21 in Healthy Volunteers.
Acronym: AMIR-21
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RNATICS GmbH (Industry)
Collaborators: LungenClinic Grosshansdorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RNATICS-2401; 2024-512351-21-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-19; First posted 2024-12-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Safety; Tolerability; Pharmacokinetics
Keywords: RCS-21; Phase I; Healthy volunteers; Inhalation
MeSH Terms: conditions — Respiratory Aspiration | interventions — Sagittal Abdominal Diameter; Saline Solution

STUDY DESIGN:
Intervention Model Description: A double blind, randomized, placebo controlled phase 1 study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single ascending dose (SAD) - Placebo (Placebo Comparator): In the single ascending dose (SAD) study, healthy volunteers receive a single inhaled dose of placebo, of the same volume as the active treatment.
  Interventions: Drug: Placebo (SAD)
- Single ascending dose (SAD) - RCS-21 (Experimental): In the single ascending dose (SAD) study, healthy volunteers will receive a single inhaled dose of 0.5 mg/participant in dose group (DG) I, 1.5 mg/participant in DG II, 4.5 mg/participant in DG III. In DG IV, the dose will be 0.5, 1.5 or 4.5 mg, depending on the safety and tolerability data obtained from DGs I-III.
  Interventions: Drug: RCS-21 (SAD)

INTERVENTIONS:
Drug: Placebo (SAD) — Inhalation of a single dose.
  Other Names: 0.9% saline solution
  Arms: Single ascending dose (SAD) - Placebo
Drug: RCS-21 (SAD) — Inhalation of a single dose.
  Arms: Single ascending dose (SAD) - RCS-21

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of RCS-21 in healthy volunteers. Participants will be asked to inhale a single dose of RCS-21 and their health status will be constantly monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Male or female aged 18 to 64 years (inclusive).
3. Women will be considered for inclusion if they are:

   * Not pregnant, as confirmed by pregnancy test (see assess- ment schedule), and not breastfeeding. AND
   * WOCBP must use one of the following highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly

     * according to recommendations by the European Heads of Medicines Agencies - from at least 14 days before the first administration of study medication until 30 days after the last administration of study medication:

       * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

         * oral
         * intravaginal
         * transdermal
       * progestogen-only hormonal contraception associated with inhibition of ovulation:

         * oral
         * injectable
         * implantable
       * intrauterine device (IUD)
       * intrauterine hormone-releasing system (IUS)
       * bilateral tubal occlusion
       * vasectomized partner (provided that this partner is the sole sexual partner of the WOCBP participant and that the vasectomized partner has received medical as- sessment of the surgical success)
       * sexual abstinence (defined as refraining from hetero- sexual intercourse during the entire study period, be- ginning 2 weeks prior to the screening visit) OR
   * Of non-childbearing potential defined according to the Clinical Trial Facilitation Group (CTFG) document "Recommendations related to contraception and pregnancy testing in clinical trials"
4. Male participants with female partner(s) of childbearing potential are eligible to participate in the study if they agree to the following during treatment and until 30 days after the last administra- tion of study medication:

   * Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator.
   * Male participants are required to use a condom during treatment and until 30 days after the last administration of study medication.
   * Female partners of male participants who have not undergone a vasectomy with the absence of sperm confirmed or a bilateral orchiectomy should consider use of effective methods of contraception during treatment and until 30 days after the last administration of study medication.
   * Sperm donation is not allowed during treatment and until 30 days after the last administration of study medication.
5. Healthy participants according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs, 12-lead Electrocardiogram (ECG), pulmonary function testing and clinical laboratory tests.
6. Body Mass Index (BMI) of 18.5 to 31.9 kg/m2 (inclusive).
7. Ability to inhale in an appropriate manner (e.g. as confirmed in the inhalation training using the PARI eFlow® device with a pla- cebo medication at the screening visit).
8. Non-smokers (including e-cigarette) or ex-smokers (with less than 10 pack years and stopped smoking for at least 5 years prior to screening visit).
9. Normal pulmonary function with Forced Expiratory Volume in the first second (FEV1) ≥ 80 % of predicted normal at screening visit. Calculations will be based on the Global Lung Function Initiative (GLI 2012) formula.

Exclusion Criteria:

1. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs, lung function or ECG at screening visit, which, in the opinion of the investigator, may either put the participant at risk because of participation in the study or may influence the results of the study, or the participant's ability to participate in the study.
2. Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, he- patic disease (asymptomatic Gilbert syndrome is allowed), renal disease, hematological disease, neurological disease, endo- crine disease (stable and asymptomatic hypothyroidism with or without Hormone Replacement Therapy (HRT) is allowed) or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
3. Having received any vaccination within the last 2 weeks before the first screening visit.
4. History or current evidence of clinically relevant allergies or idiosyncrasy to any drug or food.
5. History of allergic reactions to any active or inactive component of the study medication (including medication for bronchoscopy, e.g. salbutamol, lidocaine, midazolam or propofol).
6. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm).
7. Proneness to orthostatic dysregulation, fainting, or blackouts.
8. History or presence of any malignancy except for basalioma.
9. Chronic or acute infections or history of an acute infection during the four weeks before the first screening visit.
10. Positive results in any of the following virology tests: human im- munodeficiency virus (HIV) antibodies and antigen, Anti-hepati- tis B-core antibody (HBc-Ab), hepatitis B-surface antigen (HBs- Ag) and anti-hepatitis C virus antibody (HCV-Ab).
11. Positive drug screen (amphetamines, barbiturates, benzodiaze- pines, cannabinoids, cocaine, methadone, methamphetamine, opiates, phencyclidine, or tricyclic antidepressants).
12. History of previous administration of any registered or investiga- tional oligonucleotide-based drug.
13. History or presence of alcohol or drug abuse.
14. Use of any medication (including over-the-counter medication, herbal products) except allowed concomitant medication within 2 weeks (for biologics: 6 months) before administration of IMP or within < 10 times the elimination half-life of the respective drug, or the duration of the pharmacodynamic effect, whatever is longer.
15. Positive breath alcohol test.
16. Planned donation of oocytes, blood, organs, bone marrow dur- ing the course of the study or within 6 months after the last screening visit.
17. Participation in another clinical study with an investigational drug or device within the last 3 months or during the course of the study. For biologics, the minimum exclusion period is at least 6 months or the time of duration of the pharmacodynamic effect or 10 times the half-life of the respective drug whatever is longer before inclusion in this study.
18. Blood donation of more than 250 ml within the last 30 days before the first screening visit.
19. Anticipated non-availability for study visits/procedures.
20. Anticipated lack of willingness or inability to cooperate adequately.
21. Vulnerable participants, except WOCBP.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
SAD: Frequency and severity of AEs, frequency and severity of ARs. | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
SAD: Cmax (maximum observed plasma concentration) | up to 3 days after dosing
SAD: tmax (time of Cmax after dosing) | up to 3 days after dosing
SAD: AUC0-t last (area under the time course of the plasma concentrations up to the last quantifiable plasma concentration) | up to 3 days after dosing
SAD: AUC0-24 (area under the time course of the plasma concentrations up to 24 h after dosing, i.e. over the course of the intended dosage interval for future repeated dosing) | up to 24 h after dosing
SAD: AUC0-inf (total area under the time course of the analyte in plasma concentrations extrapolated to infinity) | up to 3 days after dosing
SAD: AUC extrapolated (relative extent of extrapolation) | up to 3 days after dosing
SAD: t½ (apparent terminal disposition half-life) and lz (apparent terminal elimination rate constant) | up to 3 days after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine (ITEM), Hanover, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participants' data that underlie the results reported in a research article will be available to researchers upon request up to 5 years after publication. Interested researchers must submit a methodologically sound proposal to amir-21@rnatics.com. Proposals will be reviewed by the sponsor to ensure that they comply with confidentiality obligations. Data will be made available within 3 months of approval of the proposal in a deidentified format in accordance with applicable privacy laws, data protection standards and consent requirements. Data requestors will need to sign a data access agreement and data will be made available through a dedicated platform.
Time Frame: The data will be available for 5 years after publication.
Access Criteria: Interested researchers must submit a methodologically sound proposal to amir-21@rnatics.com. Proposals will be reviewed by the sponsor to ensure that they comply with confidentiality obligations. Data will be made available within 3 months of approval of the proposal in a deidentified format in accordance with applicable privacy laws, data protection standards and consent requirements. Data requestors will need to sign a data access agreement and data will be made available through a dedicated platform.

REFERENCES:
- [Background] Beck C, Ramanujam D, Vaccarello P, Widenmeyer F, Feuerherd M, Cheng CC, Bomhard A, Abikeeva T, Schadler J, Sperhake JP, Graw M, Safi S, Hoffmann H, Staab-Weijnitz CA, Rad R, Protzer U, Frischmuth T, Engelhardt S. Trimannose-coupled antimiR-21 for macrophage-targeted inhalation treatment of acute inflammatory lung damage. Nat Commun. 2023 Jul 28;14(1):4564. doi: 10.1038/s41467-023-40185-1. PMID 37507393